CLINICAL TRIAL: NCT01540890
Title: Impairment of Sleep and Pattern of Breathing Before and After Opioid Withdrawal in Comparison to Patients Without Opioid Withdrawal
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr., Ruhr University of Bochum
Other Study IDs: Polysom2012
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Sleep Architecture Under Opioid Medication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- withdrawal: patients who undergo an opioid withdrawal
- opioids: patients on opioid medication without withdrawal
- opioid-free: patients with chronic pain without opioid medication

SUMMARY:
Main of the study is to assess the influence of high-dose opioids on the sleep architecture and patterns of breathing using non-invasive polysomnographic measurements before and after opioid withdrawal in patient who undergo opioid withdrawal independently from the present study. These data will be compared to polysomnographic data of patients under opioid treatment who do not undergo opioid withdrawal as well as to patients without opioid treatment.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 year, indication for opioid withdrawal (cohort 1), opioid intake (cohort 1 and 2)

Exclusion Criteria:

* plaster allergic reactions, opioid withdrawal (cohort 2), opioid intake (cohort 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatients with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
frequency of an abnormal apnoea-hypnoea index | 3 weeks

SECONDARY OUTCOMES:
changes of the sleep duration and architecture | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pain Medicine, Bochum, Germany